CLINICAL TRIAL: NCT05651932
Title: A Phase 1 Study of KTX-1001, an Oral, First-In-Class, Selective, and Potent MMSET Catalytic Inhibitor That Suppresses H3K36me2 in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of an MMSET Inhibitor in Patients With Relapsed and Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: K36 Therapeutics, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTX-MMSET-001; EUCTR No: 2022-500801-41-00 (Other: European Medicines Agency)
Record Dates: First submitted 2022-12-01; First posted 2022-12-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Myeloma; Myeloma Multiple
Keywords: NSD2; MMSET; WHSC1; T4;14; T(4;14); translocation; myeloma; RRMM
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; carfilzomib; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Single agent): KTX-1001 + dexamethasone (Experimental): Cohort A1 (single agent): KTX-1001 at RP2D1 + dex Cohort A2 (single agent): KTX-1001 at RP2D2 + dex
  Interventions: Drug: Cohort A1 & A2: KTX-1001
- Cohort B (Mezigdomide): KTX-1001 + Mezigdomide + dex (Experimental): Cohort B1 (Mezigdomide): KTX-1001 at RP2D1 + Mezigdomide + dex Cohort B2 (Mezigdomide):: KTX-1001 at RP2D2 + Mezigdomide + dex
  Interventions: Drug: Cohort B1 & B2: KTX-1001+Mezigdomide
- Cohort C (carfilzomib/KYPROLIS®): KTX-1001 + carfilzomib + dex (Experimental): Cohort C1 (carfilzomib/KYPROLIS®): KTX-1001 at RP2D1 + carfilzomib + dex Cohort C2 (carfilzomib/KYPROLIS®): KTX-1001 at RP2D2 + carfilzomib + dex
  Interventions: Drug: Cohort C1 & C2: KTX-1001 + Carfilzomib (KYPROLIS®)
- Cohort D (pomalidomide): KTX-1001 + pomalidomide + dex (Experimental): Cohort D (pomalidomide): KTX-1001 at RP2D1 or RP2D2 + pomalidomide + dex
  Interventions: Drug: Cohort D: KTX-1001+ pomalidomide (Pomalyst, Imnovid)

INTERVENTIONS:
Drug: Cohort A1 & A2: KTX-1001 — KTX-1001: Orally for 28 days each cycle until progression. Dexamethasone: Orally once weekly
  Other Names: KTX-1001; Dexamethasone
  Arms: Cohort A (Single agent): KTX-1001 + dexamethasone
Drug: Cohort B1 & B2: KTX-1001+Mezigdomide — Drug: KTX-1001: Orally for 28 days each cycle until progression Drug: Dexamethasone: Orally once weekly Drug: Mezigdomide Dexamethasone: Orally once weekly
  Other Names: Mezigdomide
  Arms: Cohort B (Mezigdomide): KTX-1001 + Mezigdomide + dex
Drug: Cohort C1 & C2: KTX-1001 + Carfilzomib (KYPROLIS®) — Drug: KTX-1001: Orally for 28 days each cycle until progression Drug: Dexamethasone: Orally once weekly Drug: Carfilzomib (KYPROLIS®): IV, once weekly for 3 weeks in each 28-day cycle
  Other Names: Carfilzomib (KYPROLIS®); Dexamethasone
  Arms: Cohort C (carfilzomib/KYPROLIS®): KTX-1001 + carfilzomib + dex
Drug: Cohort D: KTX-1001+ pomalidomide (Pomalyst, Imnovid) — Drug: KTX-1001: Orally for 28 days each cycle until progression Drug: Dexamethasone: Orally once a week Drug: Pomalidomide (Pomalyst, Imnovid): Orally, for 21 days in each 28-day cycle
  Other Names: Pomalidomide (Pomalyst, Imnovid); Dexamethasone
  Arms: Cohort D (pomalidomide): KTX-1001 + pomalidomide + dex

SUMMARY:
A Phase I study to evaluate the safety of a novel, orally available, selective, and potent small molecule inhibitor of the histone lysine methyl transferase MMSET (also known as NSD2/WHSC1) to prevent the dimethylation of H3K36 in adult patients with relapsed or refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation and expansion study in adult patients with RRMM.

In the dose escalation phase (Part A), patients will be evaluated for DLTs during Cycle 1 (28 days). The KTX-1001 MTD, RP2D, and schedule will be determined.

In the dose expansion phase (Part B), patients with t(4;14) will receive KTX-1001 at the RP2D alone and in combination with investigational therapy Mezigdomide or SOC therapy (dexamethasone, carfilzomib or pomalidomide) to further define safety and tolerability and provide preliminary efficacy information.

ELIGIBILITY:
Key Inclusion Criteria for Dose-Expansion:

* ≥ 18 years of age
* ECOG score ≤ 1
* Multiple myeloma (as per IMWG)

  * ≥ 3 prior lines of therapy, including a PI, an IMiD, and an anti-CD38 antibody
  * Patients must be refractory to their last prior therapy
  * Cohorts A1/A2: Patients must have exhausted available therapeutic options that are expected to provide a meaningful clinical benefit, either through disease relapse, treatment refractory disease, intolerance, or refusal of the therapy
  * t(4;14) confirmed by standard of care FISH testing
* Measurable disease, including at least 1 of the following criteria:

  * Serum M protein ≥ 0.50 g/dL (by SPEP)
  * Serum IgA ≥ 0.50 g/dL (IgA myeloma patients)
  * Urine M protein ≥ 200 mg/24 h (by UPEP)
  * sFLC involved light chain ≥ 10 mg/dL (100 mg/L) (patients with abnormal sFLC ratio)
  * Bone marrow plasma cells ≥ 30% (if only criterion for measurability)
* Agreement to enroll into the REMS program (Cohort D- pomalidomide cohort only)

Key Exclusion Criteria for Dose-Expansion:

* Treatment with the following therapies in the specified time period prior to first dose:

  * Patients in Cohorts B1 and B2 must not have received prior mezigdomide treatment
  * Carfilzomib in the immediate last prior line of therapy for patients enrolled in Cohorts C1 and C2
  * Pomalidomide in the immediate last prior line of therapy for patients enrolled in cohort D
  * Radiation, chemotherapy, immunotherapy, or any other anticancer therapy ≤ 2 weeks
  * Cellular therapies ≤ 8 weeks
  * Autologous transplant < 100 days
  * Allogenic transplant ≤ 6 months, or > 6 months with active GVHD
  * Major surgery ≤ 4 weeks
* Current plasma cell leukemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, and skin changes) syndrome, solitary bone lesion or bone lesions as the only evidence for plasma cell dyscrasia, myelodysplastic syndrome or a myeloproliferative neoplasm or light chain amyloidosis
* Active CNS disease
* Inadequate bone marrow function
* Inadequate renal, hepatic, pulmonary, and cardiac function
* Active, ongoing, or uncontrolled systemic viral, bacterial, or fungal infection. Permitted prophylactic medications, antimicrobials or antiretroviral therapies defined in protocol.
* Use of acid reducing agents and strong inhibitors or inducers of CYP3A4 within 14 days or 5 half-lives prior to first dose
* Strong CYP1A2 inhibitors for patients receiving pomalidomide (Cohort D)
* Active malignancy not related to myeloma requiring therapy within < 2 years prior to enrollment, or not in complete remission, with exceptions defined in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Determination of Recommended Phase 2 Dose (RP2D) and/or Maximum Tolerated Dose (MTD) Dose Expansion: Provide preliminary efficacy data on the antitumor effects of KTX-1001 in combination with other anti-myeloma therapy | Cycle 1 (28 days)
  Incidence of dose-limiting toxicity (DLTs), treatment-emergent adverse events (TEAEs), treatment-related AEs, and clinically significant changes in laboratory test results

SECONDARY OUTCOMES:
Disease Specific Response to KTX-1001± Combination Therapy | Duration of Study
  Objective Response Rate (ORR) Duration of Response (DOR) Progression Free Survival (PFS) Minimal Residual Disease (MRD)
  Per IMWG Consensus Criteria for Response and Minimal Residual Disease Assessment in Multiple Myeloma
Pharmacokinetics & Pharmacodynamics KTX-1001± Combination Therapy | Duration of Study
  Maximum plasma concentration (Cmax) of KTX-1001 Time to achieve Cmax (tmax) for KTX-1001 Area under the plasma concentration-time curve (AUC) for KTX-1001
Safety profile of KTX-1001± Combination Therapy | Duration of Study
  Frequency and severity of TEAEs, treatment-related AEs, and clinically significant changes in laboratory test results

CONTACTS AND LOCATIONS:
Locations (22):
- United States (13):
  - UCSF Medical Center - Hematology and Blood and Marrow Transplant Clinic, San Francisco, California
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - The Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Transplant Center - Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Atrium Health, Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas Southwestern Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
- University Health Network (UHN) - Princess Margaret Cancer Centre (Princess Margaret Hospital), Toronto, Ontario, Canada
- France (4):
  - Universitaire de Lille, Villeneuve-d'Ascq, France
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes) - Hotel-Dieu, Nantes
  - Centre Hospitalier Universitaire de Poitiers (CHU de Poitiers), Poitiers
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- Spain (4):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital ClÃ-nic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto de Investigacion Biomedica de Salamanca (IBSAL), Salamanca

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: K36 Therapeutics — https://www.k36tx.com/about-ktx-1001